CLINICAL TRIAL: NCT06857903
Title: Using Nudges to Recruit Human Subjects in Clinical & Translational Research
Brief Title: Using Nudges to Recruit for Health-Related Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kimberly Kaphingst, Professor, Department of Communication, and Director of Cancer Communication Research, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB_00153850; R01TR004245 (NIH)
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recruitment nudges (Experimental): Participants in this arm will receive recruitment materials that contain a set of behavioral nudges
  Interventions: Behavioral: Recruitment nudges
- Recruitment control (No Intervention): Participants in this arm will receive standard recruitment materials

INTERVENTIONS:
Behavioral: Recruitment nudges — Participants who in the intervention condition will receive recruitment materials that contain behavioral nudges
  Arms: Recruitment nudges

SUMMARY:
The goal of this clinical trial is to examine the effect of using behavioral nudges in recruitment into a minimal risk interview study among healthy adult volunteers.

Individuals will be randomized to receive recruitment materials that do or do not contain a set of behavioral nudges. Researchers will compare the effect on participation in an interview study (primary outcome) between these conditions.

ELIGIBILITY:
Inclusion Criteria:

English-speaking; 18 years of age or older

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Agreement to participate in an interview study | Within one month after initial outreach
  This outcome will be assessed as whether or not participants agree to participate in a minimal risk interview study after recruitment and consent procedures. The outcome will be assessed as yes or no.

SECONDARY OUTCOMES:
Engagement with outreach materials | Within one month after initial outreach
  This outcome will be assessed as whether or not participants respond to study outreach for a minimal risk interview study by clicking a link in the outreach email. The outcome will be assessed as yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kaphingst, ScD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will not share personally identifying information but will share participant sociodemographic characteristics and outcome data.
Supporting Information: ICF